CLINICAL TRIAL: NCT00434460
Title: Active Observational Study of the Adoption and Transfer of Clinical Practice Guidelines Through Education, for Ventilator Associated Pneumonia (ABATE VAP Study)
Brief Title: Study of Knowledge Translation of Clinical Practice Guidelines for Ventilator Associated Pneumonia
Acronym: ABATEVAP
Status: Completed | Type: Observational
Sponsor: Canadian Critical Care Trials Group (Other)
Collaborators: Kingston Health Sciences Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government); AstraZeneca (Industry); Bayer (Industry)
Responsible Party: Dr. John Muscedere, Kingston General Hospital, Queen's University
Other Study IDs: ABATE VAP
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator Associated Pneumonia; Knowledge Translation; Clinical Practice Guidelines; Education; Behaviour Change
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients receiving invasive mechanical ventilation > 48 hours.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Implementation of clinical practice guideline for ventilator associated pneumonia through education.

SUMMARY:
The purpose of this prospective, multicentre, time-series study is to develop, implement, refine, and evaluate a sustainable behaviour change strategy in the intensive care unit (ICU).

DETAILED DESCRIPTION:
Background:

In order to improve the care of our patients, it is necessary for research evidence to be translated into clinical practice. There are gaps in our understanding of knowledge translation (KT) and this is evident in the Intensive Care Unit (ICU), specifically as it applies to the prevention, diagnosis and treatment of ventilator-associated pneumonia (VAP). VAP is associated with a high burden of illness in the critically ill and there is an extensive amount of research evidence on this disease. It has been demonstrated that best practice as defined by research evidence is not uniformly applied to VAP. In addition, recent advances in VAP knowledge need be disseminated and implemented in order to improve patient safety and outcomes from VAP. A systematic process of knowledge transfer is crucial to translate this research into evidence-based bedside practice and the development and implementation of evidence based Clinical Practice Guidelines (CPGs) may facilitate VAP knowledge uptake. In addition, there is a need to study knowledge translation (KT) in the ICU since there is little information about optimal KT and CPG implementation strategies in this environment and efforts that are effective in other clinical areas may not result in meaningful change in the ICU.

Research Question:

What is the effect of VAP CPGs implemented by a multidisciplinary behaviour change strategy (consisting of multifaceted educational strategies led by local opinion leaders and augmented with reminders) on VAP guideline concordance and on clinical VAP outcomes in the ICU?

Research Plan:

Data will only be collected on consecutive patients mechanically ventilated for at least 48 hours. The following health care professionals will be studied to assess the behaviour change strategy for the VAP CPGs: physicians (intensivists, ICU fellows, ICU rotating residents), nurses, respiratory therapists, dieticians, physiotherapists and ICU administrators.

The study will be conducted in 3 phases:

1. Development of a behaviour change strategy consisting of three components:

   * Local opinion leader team
   * Educational strategy
   * Reminder system
2. Prospective implementation of the behaviour change strategy over a 24 month period
3. Prospective evaluation of the behaviour change strategy over a 24 month period

   * Concordance with VAP guidelines over time
   * Factors associated with VAP guideline concordance
   * Clinical VAP outcomes pre- and post-guideline implementation

ELIGIBILITY:
Inclusion Criteria:

* Age >= 17 years old
* Mechanically ventilated > 48 hours < 96 hours

Exclusion Criteria:

* Previous enrollment in the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients invasively mechanically ventilated > 48 hours in the critical care setting.
Sampling Method: Probability Sample
Enrollment: 1320 (Actual)
Dates: Start 2007-04; Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Muscedere, MD, Study Chair — Kingston General Hospital, Queen's University; Tasmin Sinuff, MD, PhD, Study Chair — Sunnybrook Health Sciences Centre, University of Toronto; Daren Heyland, MD, Principal Investigator — Kingston General Hospital, Queen's University; Deborah Cook, MD, Principal Investigator — St. Joseph's Healthcare, McMaster University; Peter Dodek, MD, Principal Investigator — St. Paul's University, University of British Columbia; Redouane Bouali, MD, Principal Investigator — The Ottawa Hospital, University of Ottawa; Sean Keenan, MD, Principal Investigator — Royal Columbian Hospital, University of British Columbia; Kevin Eva, PhD, Principal Investigator — McMaster University; Brenda Morgan, RN, Principal Investigator — London Health Sciences Centre, University of Western Ontario; Lori Hand, RRT, Principal Investigator — Hamilton Health Sciences Centre, McMaster University
Locations (11):
- Geisinger Health Centre, Temple University, Danville, Pennsylvania, United States
- Canada (10):
  - Royal Columbian Hospital, University of British Columbia, New Westminster, British Columbia
  - St. Paul Hospital, University of British Columbia, Vancouver, British Columbia
  - Vancouver Island Health Research Centre, Victoria, British Columbia
  - St. Joseph's Healthcare, McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Queen's University, Kingston, Ontario
  - The Ottawa Hospital, University of Ottawa, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, University of Toronto, Toronto, Ontario
  - William Osler Health Centre, Toronto, Ontario
  - Hotel Dieu Grace Hospital, Windsor, Ontario

REFERENCES:
- [Derived] Sinuff T, Muscedere J, Cook DJ, Dodek PM, Anderson W, Keenan SP, Wood G, Tan R, Haupt MT, Miletin M, Bouali R, Jiang X, Day AG, Overvelde J, Heyland DK; Canadian Critical Care Trials Group. Implementation of clinical practice guidelines for ventilator-associated pneumonia: a multicenter prospective study. Crit Care Med. 2013 Jan;41(1):15-23. doi: 10.1097/CCM.0b013e318265e874. PMID 23222254